CLINICAL TRIAL: NCT02180893
Title: Study of Paravertebral Block for Cardiac Surgery
Brief Title: The Use of Paravertebral Block for Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S12-02774
Record Dates: First submitted 2014-07-01; First posted 2014-07-03 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-02

CONDITIONS: Mitral Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paravertebral block (Experimental): Patient receiving a PVB prior to robotic mitral valve surgery
  Interventions: Other: Paravertebral Block
- No block (Placebo Comparator): Patients who did not receive PVB
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Other: Paravertebral Block — Paravertebral nerve block injection
  Arms: Paravertebral block
Other: Placebo Comparator — No block
  Patients who did not receive PVB
  Arms: No block

SUMMARY:
Pain after robotic cardiac surgery is a known problem and is often difficult to manage. Paravertebral nerve blocks are a proven method of pain relief following thoracotomy. A paravertebral block has been shown to provide good pain relief with minimal side effects, however, paravertebral blocks for robotic surgery have not been well studied. Currently the investigators routinely perform PVB on this patient population (of 50 MV robotic cases done between January and October 2012, 36 received paravertebral blocks with no adverse events noted). The investigators believe this should be studied further and that paravertebral blocks will reduce the amount of additional pain medication patients require in the first 24 hours after surgery, decrease intubation time and improve PACU and hospital discharge times.

DETAILED DESCRIPTION:
Pain after robotic cardiac surgery is a known problem and is often difficult to manage. Paravertebral nerve blocks are a proven method of pain relief following thoracotomy. A paravertebral block has been shown to provide good pain relief with minimal side effects, however, paravertebral blocks for robotic surgery have not been well studied. Currently we routinely perform PVB on this patient population (of 50 MV robotic cases done between January and October 2012, 36 received paravertebral blocks with no adverse events noted). We believe this should be studied further and that paravertebral blocks will reduce the amount of additional pain medication patients require in the first 24 hours after surgery, decrease intubation time and improve PACU and hospital discharge times.

ELIGIBILITY:
Inclusion Criteria:

* patients over the age of 18 years of age undergoing robotic mitral valve surgery.
* have capacity to understand and sign consent form

Exclusion Criteria:

* patients that are not candidates for paravertebral block as per ASRA guidelines (Horlocker, Reg Anesth Pain Med, 2010). In short, this includes patients taking specific anti platelet agents such as clopidigrel, anticoagulants such as heparin or low molecular weight heparin, or patients with an INR of greater than 1.5. -patients with a history of COPD or other respiratory diseases that would confound data on time to extubated will be excluded.
* Patients that with a diagnosis of chronic pain, or patients currently taking narcotics are excluded, as this would confound data on postoperative narcotic requirements.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Neuburger, MD, Principal Investigator — NYU
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

REFERENCES:
- [Background] Suri RM, Antiel RM, Burkhart HM, Huebner M, Li Z, Eton DT, Topilsky T, Sarano ME, Schaff HV. Quality of life after early mitral valve repair using conventional and robotic approaches. Ann Thorac Surg. 2012 Mar;93(3):761-9. doi: 10.1016/j.athoracsur.2011.11.062. PMID 22364970
- [Background] Lynch JJ, Mauermann WJ, Pulido JN, Rehfeldt KH, Torres NE. Use of paravertebral blockade to facilitate early extubation after minimally invasive cardiac surgery. Semin Cardiothorac Vasc Anesth. 2010 Mar;14(1):47-8. doi: 10.1177/1089253210363009. PMID 20472625

RESULTS

PARTICIPANT FLOW:
Groups:
- Paravertebral Block: Patient receiving a PVB prior to robotic mitral valce surgery
  Paravertebral Block: Paravertebral nerve block injection
- No Block: Patients who did not receive PVB
  Placebo Comparator: No block
  Patients who did not receive PVB
Period: Overall Study
Arm/Group | Paravertebral Block | No Block
Started | 30 | 30
Completed | 27 | 23
Not Completed | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paravertebral Block | No Block | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (12.2) | 62.2 (11.9) | 61.15 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 12 | 17
  Male | 25 | 18 | 43

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Fentanyl
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: microgram/kilogram
Arm/Group | Paravertebral Block | No Block
Number analyzed (Participants) | 27 | 23
microgram/kilogram | 4.51 (2.5) | 6.14 (2.88)

2. Primary Outcome: Visual Analog Scale (VAS) Pain Scores
Description: Possible scores range from 0-10, with 0 being no pain and 10 being highest level of pain
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paravertebral Block | No Block
Number analyzed (Participants) | 27 | 23
units on a scale | 3.33 (1.52) | 4.13 (1.25)

3. Secondary Outcome: Participant Satisfaction
Description: Participants were asked whether or not they were satisfied with their postoperative pain control (yes or no)
Time Frame: 48 hours
Measure: Number; unit: percentage of "yes" responders
Arm/Group | Paravertebral Block | No Block
Number analyzed (Participants) | 27 | 23
percentage of "yes" responders | 100 | 86.7

4. Secondary Outcome: Participant Satisfaction Score
Description: Participants were asked to score their satisfaction with their postoperative pain control on a scale of 0 (least satisfied) to 10 (most satisfied)
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paravertebral Block | No Block
Number analyzed (Participants) | 27 | 23
units on a scale | 8.44 (1.25) | 6.83 (1.90)

ADVERSE EVENTS:
Arm/Group | Paravertebral Block | No Block
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes